CLINICAL TRIAL: NCT05351177
Title: The Feasibility of an 8-Week High-Intensity Interval Training (HIIT) or Concurrent Training (CT) Programme in Overweight and Obese Adult Males
Brief Title: 8-Weeks of High-Intensity Interval Training or Concurrent Training in Overweight and Obese Adult Males
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sunderland (Other)
Responsible Party: Principal Investigator, Jordan Bell, PhD Researcher, University of Sunderland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 009112
Record Dates: First submitted 2022-04-08; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Interval Training Group (Experimental): Participants in the High-Intensity Interval Training (HIIT) group will complete 8 weeks of twice-weekly HIIT of 30 minutes in duration. Heart rate, ratings of perceived exertion, affect and enjoyment will be assessed. This will include a five minute warm-up on a cycle ergometer, followed by 10 x 60 second repetitions on the cycle ergometer interspersed with 60 seconds rest. A five minute cooldown will follow on the cycle ergometer.
  Interventions: Other: Exercise Training
- Concurrent Training Group (Experimental): Participants in the Concurrent Training (CT) group will complete 8 weeks of twice-weekly CT of 30 minutes in duration. Heart rate, ratings of perceived exertion, affect and enjoyment will be assessed. This will include a five minute warm-up on a cycle ergometer, followed by two sets of four then eight repetitions of deadlift, squat, bench press and shoulder press resistance exercises. Thereafter, 5 x 60 second HIIT cycling intervals will be completed on a cycle ergometer, after which a five minute cooldown will ensue.
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — Either of; 8-weeks twice-weekly High-Intensity Interval Training or Same-Session Concurrent Exercise Training.

SUMMARY:
Overweight and obesity is becoming increasingly prevalent, constituting 64% of all adults in England, causing an incessant rise in cost to the National Health Service. Exercise and physical activity have the potential to reduce incidence of overweight and obesity, as well as improve obesity-related ill health. However, overweight and obese individuals are inherently sedentary and do not meet exercise guidelines. Same-session concurrent exercise training may be the most efficient exercise strategy to incorporate both cardiovascular- and strength-based exercise, both of which are vital for health-related benefits. This research project will aim to determine the feasibility of completing an 8-week concurrent exercise training programme in overweight and obese sedentary males. This study will aim to recruit adult males with a BMI above 25 kg.m2, who are otherwise healthy, but not regularly achieving exercise guidelines (less than 150 minutes of physical activity and 2 strength training sessions per week). Participants will undergo baseline and post-training testing of cardiorespiratory fitness, strength, heart and metabolic health, as well as a series of questionnaires and a semi-structured interview. They will then be randomised into one of two groups (high-intensity interval training or concurrent training) to complete twice-weekly exercise sessions for 8 weeks. The aims of this study are to evaluate the feasibility of performing 8-weeks of either concurrent, resistance or high-intensity interval training in overweight and obese males. This will be determined through assessment of cardiorespiratory fitness, strength, heart health, metabolic health, enjoyment, adherence and attendance.

DETAILED DESCRIPTION:
This study will incorporate a randomised controlled design, involving three distinct phases for two separate groups of participants. Participants will be randomly assigned into one of four groups via a computerised randomiser (Sealed Envelope Ltd., 2020), with a 1:1 allocation ratio using block sizes of two. These groups will consist of a HIIT group and concurrent training group. Three phases will be spread across 10 weeks for each participant:

* Phase 1: baseline testing for all groups (week 1)
* Phase 2: an 8-week exercise intervention for three experimental groups (weeks 2 - 9)
* Phase 3: post-intervention testing for all groups (week 10). Participants will be provided with all of the study information and given the opportunity to ask questions from the researchers before providing informed consent. Full pre-exercise screening in accordance with the American College of Sports Medicine (ACSM) guidelines for exercise testing will be conducted. All participants will be overweight or obese (BMI > 25 kg.m2) and sedentary but will be excluded if pre-exercise screening highlights any other cardiovascular disease risk factor.

Phase One: Baseline Testing Once included in the study, participants will be randomised into one of two groups (HIIT or Concurrent). Both groups will perform exactly the same baseline testing procedures over the course of two days during Week 1 of the study duration. On the first day participants will arrive at the University of Sunderland exercise testing laboratory having completed a 12 hr fast, having abstained from caffeine and alcohol consumption for 24 hr and not exercised in the previous 72 hrs, and asked to consume 500 ml of water 1 hour prior to arrival.

Fasted blood samples will then be collected. Plasma glucose, lipid profile and HbA1C concentrations will be assessed via a fingertip capillary blood sample. Each fingertip capillary sample will be performed using a safety lancet. Blood samples will be immediately analysed and disposed of in clinical waste. Samples will be analysed via a CardioChek PA portable lipid analyser, HemoCue Hb analyser and Biosen blood glucose analyser. Once sterilised with an alcohol wipe, skin perforations will only be made on the fingertips, and participants will be provided with adhesive dressings should they be requested. There will then be a short break (~30 minutes) in which participants will be provided with a light breakfast of toasted white bread (50 g) with strawberry jam (40 g), constituting a total of 75 g Carbohydrate. After consuming the breakfast participants will score their appetite via a visual analogue scale (Flint et al., 2000). The breakfast will standardise pre-exercise nutritional status both between- and within-participants.

Pre-exercise health screening will be completed in line with American college of sports medicine (ACSM) and University of Sunderland guidelines. Inclusive of this screening procedure will be anthropometric measures (height, mass, waist and hip circumference) as well as resting heart rate (determined via a Polar heart rate monitor and wristwatch) and resting blood pressure (via automatic sphygmomanometer). Participants will be excluded upon evidence of any contraindications to exercise (ACSM, 2020). In addition to this, body fat will be determined via the BodyStat 1500 bioelectrical impedance device. This will not occur if the participant has any form of pacemaker device. Hydration status will be determined prior to bioelectrical impedance via an Osmocheck portable analyser.

Participants will complete strength testing measures at the University of Sunderland exercise testing gym. Each participant will complete an 8-repetition maximum (8RM) test for each of the following exercises: barbell squat, barbell deadlift, barbell chest press, machine shoulder press under supervision of a qualified gym instructor. The protocol will follow a reliable and valid method set out by Taylor and Fletcher (2012). Participants will perform familiarisation with each exercise, finding a resistance they deem 'somewhat easy' for one repetition and practising until they demonstrate correct technique to the qualified gym instructor. Thereafter, increasing amounts of load will be added until participants can complete an 8th but not a 9th repetition using correct technique. If more than 8 repetitions can be performed the load will be increased 5 - 10%, with 3 mins rest allowed between attempts, and 5 mins between exercises. Grip strength will then be assessed in both hands via portable dynamometer. The strength tests will be the first exercise assessments completed in order to minimise influence of the interference effect (Laursen and Buchheit, 2019). This will conclude day one of baseline testing, which will take 1.5 - 2 hours to complete.

On day two participants will arrive at the University of Sunderland a minimum of 24 hrs after their first visit, having completed a 12 hr fast, no additional exercise and continued their abstinence of caffeine and alcohol the previous 72 hrs. Participants will complete an oral glucose tolerance test (OGTT) to assess insulin sensitivity and glucose uptake. Participants will consume 75 g of carbohydrate in the form of a commercially available glucose solution - a safe and standardised amount to administer (Belfiore et al., 1997). Thereafter, the participant will remain in the laboratory for 120 mins, with fingertip blood samples taken at rest and at 20 min intervals to determine plasma glucose concentrations. In total, the participant will have seven fingertip blood samples. The 20 min gaps between blood samples will be used to familiarise participants with various scales that will be used throughout the study, including ratings of perceived exertion (RPE - Borg, 1982), the physical activity enjoyment scale (PACES, Kendzierski & DeCarlo, 1991) and the feeling scale (Hardy & Rejeski, 1989). Participants will also complete the PRETIE-Q questionnaire for understanding preferences and tolerances of exercise intensity (Ekkekakis, 2005). Likewise, participants will complete a semi-structured interview with the lead researcher of ~20 minutes in duration. Questions will focus on personal barriers to regular physical activity and previous exercise experiences. The questions are based on previous research which has sought to understand amounts of physical activity completed and barriers to exercise participation (McIntosh et al., 2016; Willett et al., 2019). This interview will be recorded and transcribed, with each participant assigned a code for the duration of the study so that all information remains anonymous. The template for both baseline and post-intervention interviews are included in attachments.

Participants will then complete a cardiopulmonary exercise test (CPET) in the exercise testing laboratory. A 12-lead electrocardiograph (ECG) with the Mason-Likar electrode placement will be taken at rest and throughout exercise. Participants will complete the CPET on a Lode cycle ergometer, involving a 5 min warm-up at 60 W to prevent musculoskeletal injury and a ramped workload protocol (individualised 15 - 25 W.min-1) that will terminate at volitional exhaustion (8 - 12 mins). Respiratory gases will be collected with breath-by-breath measurements via a metalyzer (Cortex, Metalyzer) and converted to 30 second averages for ease of analysis. The highest volume of oxygen (VO2) value attained during the test when converted to 30 second averages will be used as the participants VO2peak. The anaerobic threshold (AT) will be identified as the point at which the ventilatory rate (Ve) and volume of carbon dioxide (VCO2) break linearity with the volume of oxygen (VO2), using the v-slope method (Wasserman, 1986) from the middle 5 of 7 breath-by-breath average. After the CPET participants will undergo a 5-minute unloaded cool down during which cardiovascular measures will continue to be monitored. This will conclude day two of baseline testing, with the visit totalling ~3 hours in duration.

Participants will also undergo a standard transthoracic echocardiogram (TTE) to determine structural cardiac adaptations. An initial assessment will be performed at the University of Sunderland in the school of medicine, lasting no longer than 30 minutes. A second assessment will be completed at the end of the training programme. A series of echocardiographic parameters will be obtained, including wall thickness, ventricular ejection fraction and left ventricular mass. The screening will be carried out by a qualified cardiac physiologist. Participants will be immediately excluded from the study with the presence of any cardiac abnormalities and referred to their general practitioner. The TTE may take place on either day of testing measures, depending on availability of the cardiologist and/or echocardiogram at the University of Sunderland. Participants will be notified prior to their arrival on which day their TTE will take place.

In addition, throughout the baseline testing week habitual diet and physical activity levels will be recorded. A representative 3 - 4 day period will be selected in which a diet diary will be self-reported by all participants, with each instructed on how this should be completed. Two weekdays as well as one weekend day will be completed as a minimum. This will be analysed for energy intake and relative macronutrient intakes by the researchers. Habitual physical activity levels will be assessed via ActiGraph wGT3X-BT (ActiGraph, USA) activity monitors. Each participant will be instructed on how to correctly place the monitor around the waist, which will be in place for 3 - 5 days across the week of baseline testing (a minimum of one midweek, and both Saturday and Sunday). The raw accelerometer data will be uploaded to Actilife Software (ActiGraph, USA), from which energy expenditure and time spent in moderate to vigorous exercise will be extracted.

Phase 2: Exercise Interventions Three groups will undergo a twice-weekly, 8-week exercise training programme. Each exercise session will be separated by a minimum of 48 hrs to aid recovery, prevent incidence of musculoskeletal injury and standardise the programme.

HIIT Group Participants in the HIIT group will arrive at the exercise testing laboratory at the University of Sunderland for each visit. Resting measures of heart rate and blood pressure will be collected. The HIIT protocol will be completed on a Lode cycle ergometer, with a 5 min warm-up at 60 W followed by a stretching period to prevent musculoskeletal injury. The protocol will follow a modified-style HIIT design with 10 x 60 s intervals interspersed with 60 s rest. The intensity of the HIIT intervals will be set using the delta (Δ) method in order to create individualised workloads specific to the participant, ensuring workloads are well matched for all individuals. This will involve setting the intensity of exercise based on each participant's CPET results, using the workload at the AT, the VO2peak and a percentage of the gap between these two. All participants will cycle at 80% Δ for 60 s followed by 60 s rest, for a total of 20 minutes. Following the final HIIT interval participants will continue cycling for 5 min at 60 W in a cooldown phase. This will constitute a total session duration of 30 mins. All HIIT sessions will be supervised by a member of the research team.

Concurrent Group Participants in the same-session concurrent training group will perform training sessions that involve 50% of the HIIT and Resistance protocols. Participants will arrive at the exercise testing laboratory and gym at the University of Sunderland for each visit. Resting measures of heart rate and blood pressure will be collected. Participants will complete a 5 min cycling warm-up at 60 W on a cycle ergometer followed by a stretching period. The resistance training component will be completed first and on the same four exercises as baseline testing in order to minimise influence of the interference effect. However, participants will only complete 4 repetitions of their 8RM, be given 30 s rest and then complete 1 set of 8 repetitions at 100% of their 8RM, with 60 s rest before moving on to the next exercise. This will ensure 150 s is spent on each exercise, allowing for a total of 10-minutes on resistance exercises. Participants will then move onto the Lode cycle ergometer to complete the HIIT aspect of their training session. They will complete 5 x 60 s intervals at 80% Δ interspersed with 60 s rest, completing a total of 10 mins of HIIT. A 5 min cycling cooldown on the Lode cycle ergometer at 60 W will be completed in the same manner as the other groups. This will ensure that the concurrent training session will last 30 mins in duration. All concurrent sessions will be supervised by a member of the research team and a qualified gym instructor.

For all three groups participants will be fitted with Polar Bluetooth heart rate monitors for continuous measurement throughout exercise. Five minutes after the end of the exercise session participants will be asked to complete a session-rating of perceived exertion (CR100 Scale), the PACES enjoyment scale and the Feeling Scale. In the first, fourth and eighth weeks, one of the training sessions will be used to collect additional data on the physiological load across the programme. The HIIT group will have respiratory gases analysed during their workout, the resistance group will have a post-exercise fingertip capillary blood sample to determine lactate concentration via Lactate Pro 2 (Arkray, Japan). The concurrent group will have both respiratory gases and lactate concentration assessed after the resistance and HIIT aspects respectively.

Phase 3: Post-intervention Testing Post-intervention testing will be completed by all groups and replicate all of the tests that took place across two days during baseline testing. The only change from these tests will be that the semi-structured interview will focus on the overall experience of the training intervention, the participant's desire to continue and the feasibility of employing such an exercise intervention in free-living conditions. There would not be a post-exercise semi-structured interview for any participants in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult males (18 - 66 years)
* Overweight or obese ( >25 kg.m2 body mass index - BMI)
* Normally achieve less than 150 minutes of moderate-intensity or 75 minutes of vigorous-intensity physical activity and 2 strength training sessions per week
* No existing comorbidities (e.g. type 2 diabetes mellitus, hypertension)
* Have not completed an exercise training programme in the previous 3 months
* Are not currently completing a weight loss intervention (e.g. pharmacological/dietary)
* No existing musculoskeletal injury
* Have not tested positive for COVID-19 within the previous 6 months and are asymptomatic from COVID-19 related symptoms.
* Have adverse or allergic reactions to the allergens present in white bread or strawberry jam (e.g. Gluten).

Ages: 18 Years to 66 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Adherence | Throughout intervention (8 weeks)
  Feasibility of the study will be measured via adherence to the exercise programme (number of intervals of HIIT or repetitions of resistance exercises completed).
Attendance | Throughout Intervention (8 weeks)
  Number of exercise training sessions attended.
Enjoyment | Throughout intervention (8 weeks)
  Scores will be taken from the Physical Activity Enjoyment Scale (PACES), which will be completed at the end of each exercise session.
In-Session Heart Rate | Throughout intervention (8 weeks)
  The heart rate (in beats per minute) at the end of each HIIT interval or set of resistance exercise measured via Polar Wristwatch.
Ratings of Perceived Exertion | Throughout intervention (8 weeks)
  The Rating of Perceived Exertion (RPE) at the end of each HIIT interval or resistance exercise, provided by each participant on the Borg category-ratio 100 scale, expressed in arbitrary units.

SECONDARY OUTCOMES:
Body Mass | Pre and Post (Weeks 1 and 10)
  Measured in kilograms to the nearest 0.1kg, from standing scales, with participants barefoot and stripped to shorts and t-shirt.
Height | Pre and Post (Weeks 1 and 10)
  Taken via stadiometer with participants stood barefoot and positioned with their heels facing toward the stadiometer, standing upright with their shoulders back and face forward in the Frankfurt plane. Height was taken to the nearest 0.1 cm from the vertex
Waist Circumference | Pre and Post (Weeks 1 and 10)
  Measured by tape measure to the nearest 0.1 cm when placed directly on the skin, in the horizontal plane midway between the lowest rib and the iliac crest.
Hip Circumference | Pre and Post (Weeks 1 and 10)
  Measured by tape measure to the nearest 0.1 cm when placed directly on the skin, in the horizontal plane at the maximum posterior extension of the buttocks
Body Fat | Pre and Post (Weeks 1 and 10)
  Determined via bioelectrical impedance and reported as a percentage with participants requested to consume 400 ml water 1 hour prior to their visit. Participants remained in a supine position, with electrodes affixed to their right wrist and ankle.
Body Mass Index | Pre and Post (Weeks 1 and 10)
  Product of height and body mass expressed in kg/m2.
VO2Peak | Pre and Post (Weeks 1 and 10)
  The maximum oxygen uptake value achieved during an incremental cardiopulmonary exercise test, determined via online gas-analysis through breath-by-breath measurements and expressed in ml/kg/min-1.
Left Ventricular Volume | Pre and Post (Weeks 1 and 10)
  Measured via echocardiogram, in both systole and diastole as well as two- and four-chamber views, expressed in ml.
Left Ventricle | Pre and Post (Weeks 1 and 10)
  Size measured via echocardiogram during diastole in cm.
Ejection Fraction | Pre and Post (Weeks 1 and 10)
  Measured via echocardiogram as a product of the end systolic minus end diastolic volumes and expressed as a percentage.
Fasting Plasma Glucose | Pre and Post (Weeks 1 and 10)
  Fasting plasma glucose concentration measured in mmol/L via fingertip capillary blood sample and portable glucose analyser.
Low-Density-Lipoprotein Concentration | Pre and Post (Weeks 1 and 10)
  Low-Density-Lipoprotein (LDL) concentration in mmol/L determined via fingertip capillary blood sample and portable analyser.
High-Density-Lipoprotein Concentration | Pre and Post (Weeks 1 and 10)
  High-Density-Lipoprotein (HDL) concentration in mmol/L determined via fingertip capillary blood sample and portable analyser.
Cholesterol | Pre and Post (Weeks 1 and 10)
  Total cholesterol concentration in mmol/L determined via fingertip capillary blood sample and portable analyser.
Triglycerides | Pre and Post (Weeks 1 and 10)
  Serum triglyceride concentration in mmol/L determined via fingertip capillary blood sample and portable analyser.
HbA1C | Pre and Post (Weeks 1 and 10)
  HbA1C concentration in mmol/mol determined via fingertip capillary blood sample and portable analyser.
Area Under the Glucose Curve | Pre and Post (Weeks 1 and 10)
  The Area Under the Curve (AUC) from an Oral Glucose Tolerance Test (OGTT) after consumption of a 75g Glucose solution and measurements of plasma glucose concentration at 20-minute intervals for 120 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sunderland, Sunderland, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No